CLINICAL TRIAL: NCT07298551
Title: Construction of an Assessment Model for Vitiligo Disease Activity and Treatment Prognosis Based on Peripheral Blood Cytokine Profiles
Brief Title: Building an Assessment Model for Vitiligo Activity and Prognosis Using Peripheral Blood Cytokine Profiles
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJPF-LCY-V2025113
Record Dates: First submitted 2025-12-08; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy people
  Interventions: Diagnostic Test: Serum Cytokine Assay
- vitiligo patients: Vitiligo patients were assigned to one of the following treatment groups based on clinical protocols: topical therapy group, systemic therapy group, phototherapy group, or combination therapy group.
  Interventions: Diagnostic Test: Serum Cytokine Assay

INTERVENTIONS:
Diagnostic Test: Serum Cytokine Assay — Detect the expression levels of cytokines including IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-17, IFN-α, IFN-γ, and TNF-α in peripheral blood.

SUMMARY:
Vitiligo is a chronic autoimmune disorder characterized by depigmented patches on the skin, which can pose significant psychosocial challenges, particularly for individuals with darker skin tones. Compared to the general population, individuals with vitiligo are more likely to experience immune-mediated diseases or psychological comorbidities. Studies confirm that the combined prevalence of depression and anxiety among vitiligo patients reaches 8% and 35.8%, respectively. Notably, the anxiety prevalence rate is comparable to that seen in other severely debilitating skin conditions such as eczema and psoriasis. However, the progression, stability, and recurrence of vitiligo exhibit high unpredictability. Unlike other inflammatory skin diseases such as psoriasis or atopic dermatitis, there is currently a lack of objective, sensitive biological markers in clinical practice to predict disease activity, forecast treatment response, or assess long-term prognosis. Decisions primarily rely on the attending physician's assessment of disease activity, affected areas, severity, and repigmentation potential. Furthermore, clinical signs of active vitiligo are only observable in some active-phase patients, introducing delays and subjectivity. This leads to reactive treatment decisions, increasing the likelihood of missing the optimal intervention window. Cytokines are small-molecule polypeptides or glycoproteins synthesized and secreted by the body's cells, possessing diverse biological activities. They play a central role in physiological and pathological processes such as immune regulation, anti-infection, and anti-tumor responses. The "Twelve Cytokine Panel" is a clinical test utilizing advanced flow cytometry for the combined analysis of 12 core cytokines. The cytokines included in this test are IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-17, IFN-α, IFN-γ, and TNF-α. This panel comprehensively reflects innate immune and T-cell immune responses, providing crucial laboratory evidence for evaluating the functional status of the immune system and inflammatory network. Cytokines serve as core messenger molecules in the autoimmune pathogenesis of vitiligo, forming a complex inflammatory network that governs the entire process of immune attacks against melanocytes. Consequently, detecting specific cytokine profiles not only deepens our understanding of vitiligo's disease mechanisms but also holds immense potential clinical value in assessing disease activity, monitoring treatment efficacy, and developing novel targeted therapies.

DETAILED DESCRIPTION:
Background: Pigmentary skin disorders constitute a group of conditions characterized by the loss of normal pigmentation in the skin and/or mucous membranes. Currently, there is a lack of objective, sensitive biological markers in clinical practice to predict disease activity, forecast treatment response, and assess long-term prognosis. Diagnosis primarily relies on the attending physician's evaluation of disease activity, affected areas, severity, and repigmentation potential. Furthermore, clinical signs of active vitiligo are only observable in some active-phase patients, leading to delayed and subjective assessments. This results in passive treatment decisions and increases the likelihood of missing the optimal intervention window. The "Twelve Cytokine Panel" is a clinical test utilizing advanced flow cytometry for the combined analysis of 12 core cytokines. The cytokines included in this test are Interleukin-1β (IL-1β), Interleukin-2 (IL-2), Interleukin-4 (IL-4), Interleukin-5 (IL-5), Interleukin-6 (IL-6), Interleukin-8 (IL-8, also known as CXCL8), Interleukin-10 (IL-10), Interleukin-12p70 (IL-12p70), Interleukin-17 (IL-17), Interferon-alpha (IFN-α), Interferon-gamma (IFN-γ), and Tumor Necrosis Factor-alpha (TNF-α). This comprehensive assessment reflects innate immune and T-cell immune responses, providing crucial laboratory evidence for evaluating immune system and inflammatory network function. Study Design: Based on this research context, peripheral blood samples were collected from 100 vitiligo patients and 25 healthy controls to measure cytokine levels. The vitiligo patient group was stratified according to clinical treatment modalities. Changes in peripheral blood cytokine levels were tracked at 1-month and 6-month treatment follow-ups, compared against cytokine levels in healthy controls, and correlated with clinical repigmentation status and psychological treatment efficacy. This approach aims to predict vitiligo progression and prognosis through serum inflammatory cytokine levels, thereby enhancing the formulation of clinical treatment strategies. Statistical Methods: Data will undergo statistical inference using chi-square tests, Wilcoxon signed-rank tests, Kruskal-Wallis H tests, Dunn's multiple comparison tests, Pearson correlation analysis, and logistic regression (significance: p ≤ 0.05). Ethics and Compliance: Approved by the Ethics Committee of the First Affiliated Hospital of Air Force Medical University. Informed consent must be obtained from all participants' guardians.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically confirmed vitiligo (diagnosis criteria refer to the Consensus on Vitiligo Diagnosis and Treatment (2018 Edition) established by the Pigment Disorders Group of the Dermatology and Venereology Professional Committee of the Chinese Association of Integrative Medicine) and a healthy control group.
* Aged 18 years or older, no gender restrictions
* Possess an elementary school education or higher
* Voluntarily participate in this study

Exclusion Criteria:

* Patients who have used antibiotics, corticosteroids, or immunosuppressants within the past month
* Patients with severe cardiovascular or cerebrovascular disease, severe diabetes, severe infection, or other major illnesses resulting in poor physical condition
* Patients with photosensitive disorders, skin tumors, autoimmune diseases, or hematological disorders
* Pregnant or lactating women
* Patients with poor psychological stability or compliance who cannot cooperate with follow-up visits or nursing care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult participants aged 18 or older, divided into a case group of clinically confirmed vitiligo patients and a healthy control group, all possessing at least an elementary school education and voluntarily participating. Excluded are individuals who have recently used antibiotics, corticosteroids, or immunosuppressants; those with significant comorbidities such as severe cardiovascular disease, diabetes, infections, photosensitive disorders, skin tumors, autoimmune or hematological diseases; pregnant or lactating women; and those with psychological or compliance issues that would hinder follow-up or care cooperation.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Achieving T-VASI 50 | "Baseline""4 week""24 week"
  The proportion of patients achieving a 50% or greater improvement from baseline in the Total Vitiligo Area Scoring Index
Proportion of Patients Achieving F-VASI 75 | "Baseline""4 week""24 week"
  The proportion of patients achieving a 75% or greater improvement from baseline in the Facial Vitiligo Area Scoring Index

SECONDARY OUTCOMES:
Vitiligo Quality of Life Instrument | "Baseline""4 week""24 week"
  Acronym: VitiQoL
  Description & Structure: The VitiQoL is a 15-item, disease-specific quality of life questionnaire designed for patients with vitiligo. It comprises three subdomains: Psychological Burden, Activity Limitation, and Appearance Concerns. Patients are asked to recall their experience over the past week and rate how bothered they have been by each item on a 5-point Likert scale (0 = "Never", 1 = "Rarely", 2 = "Sometimes", 3 = "Often", 4 = "Always").
  Scoring Range: The total score ranges from 0 to 60, calculated by summing the scores of all 15 items.
  Score Direction & Interpretation: A higher total score indicates greater impairment in disease-specific quality of life (worse outcome). A decrease in score from baseline represents an improvement.
Chinese Vitiligo Quality of Life Scale | "Baseline""4 week""24 week"
  Acronym: CVQLS
  Description: The CVQLS is a 25-item questionnaire developed specifically for Chinese vitiligo patients. It assesses disease impact over the past month across three dimensions: Daily Life Restriction, Disease Burden, and Social Limitation. Items are scored from 0 ("Not at all") to 4 ("Extremely").
  Scoring Range: 0 to 100. The total score is the sum of all item scores.
  Score Interpretation: A higher score indicates worse quality of life (greater impairment). A decrease in score represents improvement.
  Rationale: Selected for cultural relevance to Chinese patients, addressing concerns like economic burden and social stigma not fully captured by international tools.
Hospital Anxiety and Depression Scale | "Baseline""4 week""24 week"
  Acronym: HADS
  Description & Structure: The HADS is a 14-item self-assessment scale designed to screen for states of anxiety and depression in non-psychiatric hospital settings. It consists of two independent subscales: the Anxiety subscale (HADS-A) and the Depression subscale (HADS-D), each containing 7 items. Each item is scored on a 4-point scale (0-3) reflecting the frequency of symptoms over the past week.
  Scoring Range:
  HADS-Anxiety (HADS-A) subscale score: 0 to 21.
  HADS-Depression (HADS-D) subscale score: 0 to 21.
  *(Note: A total HADS score [0-42] is not recommended for primary interpretation as it combines distinct constructs.)*
  Score Direction & Interpretation: A higher score on either subscale indicates a greater severity of anxiety or depressive symptoms (worse outcome).
  Clinical Cut-off Reference (per subscale): Scores of 0-7 are generally regarded as being in the normal range, 8-10 as borderline/mild, 11-14 as moderate, and 15-21 as severe.
Serum cytokine concentrations | "Baseline""4 week""24 week"
  Expression levels of cytokines including IL-1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-17, IFN-α, IFN-γ, and TNF-α in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: Undecided